CLINICAL TRIAL: NCT06250712
Title: Hativ® ELectrocardiogram Monitoring on Patients With Suspected Arrhythmia
Acronym: HELP-A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Young Jun Park, Assistant Professor, Wonju Severance Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CR223024
Record Dates: First submitted 2024-01-31; First posted 2024-02-09 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-08

CONDITIONS: Arrhythmia
Keywords: Palpitation; Dizziness; Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac; Dizziness

STUDY DESIGN:
Intervention Model Description: In the 588 patients who require additional testing due to arrhythmia symptoms, continuous single lead ECG or intermittent handheld ECG will be randomly assigned to the test for 1 month. If arrhythmia symptoms are not diagnosed after 1 month, cross over the device and use it for another month for evaluation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continous ECG Patch (Experimental): In this arm, continuous patch ECG was used.
  Interventions: Device: Continous ECG Patch
- Intermittent handheld ECG (Active Comparator): In this arm, intermittent handheld ECG was used.
  Interventions: Device: Intermittent handheld ECG

INTERVENTIONS:
Device: Continous ECG Patch — Using a continuous patch ECG for 1 week during 1 month
  Arms: Continous ECG Patch
Device: Intermittent handheld ECG — Using a handheld ECG twice daily and when symptoms are present during 1 month
  Arms: Intermittent handheld ECG

SUMMARY:
HELP-A study is a single-center, randomized, controlled trial. A total of 588 patients enrolled during the 2 years of enrollment period and followed for 1 month of follow-up period. This study aims to compare diagnostic yield between continuous ECG Patch and intermittent handheld ECG in patients with arrhythmia symptoms.

DETAILED DESCRIPTION:
HELP-A study is a single-center, randomized, controlled trial designed to compare diagnostic yield, arrhythmia detection rate, user convenience, and cost-effectiveness between continuous ECG Patch and intermittent handheld ECG in patients with arrhythmia symptoms. Patients who have symptoms of arrhythmia but are not diagnosed on a 12-lead ECG and require additional tests. A total of 588 patients enrolled during the 2 years of enrollment period and followed for 3 month of follow-up period. Patients will be assigned to continuous patch ECG or intermittent handheld ECG and will be examined for one month. If there is no diagnosis after a month, the patient will be crossed over to another device and examined for another month.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have arrhythmia symptoms but are not diagnosed on a 12-lead electrocardiogram and require additional tests.
* Patients who can use a smartphone

Exclusion Criteria:

* Patients who have cardiac implantable electronic devices(CIEDs)
* Patients who can't use handheld ECG

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 1 month
  (Number of patient with triggered event without arrhythmia + Number of patients with clnically significant arrhytmia) / total patients

SECONDARY OUTCOMES:
Arrhythmia detection rate | 3 month
  Compare the arrhythmia diagnosis rate between the two devices.
Cost-effectiveness | 3 month
  Compare Total medical cost incurred for arrhythmia symptoms between the two devices
Chagne of Quality of Life | Baseline, 3 month
  Compare Quality Of Life using Euro QOL-5D-5L between the two devices
User convenience | 3 month
  Comparison of User convenience using questionnaires in patients who used both devices (ease, portability, satisfaction, etc.) The questionnaire consists of 5 scales from 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Young Jun Park, MD, Principal Investigator — Wonju Severance Christian Hopsital
Locations (3):
- South Korea (3):
  - Chonnam National University Hospital, Gwangju, Dong-gu Jaebongro 42
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do, Hwaseong-si Keunjaebong-gil 7

REFERENCES:
- [Background] Raviele A, Giada F, Bergfeldt L, Blanc JJ, Blomstrom-Lundqvist C, Mont L, Morgan JM, Raatikainen MJ, Steinbeck G, Viskin S, Kirchhof P, Braunschweig F, Borggrefe M, Hocini M, Della Bella P, Shah DC; European Heart Rhythm Association. Management of patients with palpitations: a position paper from the European Heart Rhythm Association. Europace. 2011 Jul;13(7):920-34. doi: 10.1093/europace/eur130. No abstract available. PMID 21697315
- [Background] Turnbull S, Garikapati K, Bennett RG, Campbell TG, Kotake Y, Mahajan R, Marschner S, Byth K, Chow CK, Kumar S. Utility of a Handheld, Single-Lead ECG Device for Diagnosis of Cardiac Arrhythmias. J Am Coll Cardiol. 2023 Jun 13;81(23):2292-2294. doi: 10.1016/j.jacc.2023.03.428. No abstract available. PMID 37286259
- [Background] Schreiber D, Sattar A, Drigalla D, Higgins S. Ambulatory cardiac monitoring for discharged emergency department patients with possible cardiac arrhythmias. West J Emerg Med. 2014 Mar;15(2):194-8. doi: 10.5811/westjem.2013.11.18973. PMID 24672611